CLINICAL TRIAL: NCT06018064
Title: Investigating the Fit and Satisfaction of an Innovative Device - Prone to Excellence: A Tummy Time Device Prone Positioner for Infants With Medical Complexities Including Artificial Airways: A Design Pilot Study
Brief Title: Investigating Fit and Satisfaction of the Prone Positioner
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Brandi Dorton, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002288
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Infant Development

STUDY DESIGN:
Intervention Model Description: Infants between the ages >44 weeks gestational age to 18 months of age with complex medical conditions, particularly those with tracheostomies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): Subjects who are placed in the Prone Positioner for evaluation
  Interventions: Device: Prone Positioner

INTERVENTIONS:
Device: Prone Positioner — An innovative device to allow for infants to be supported while in the prone position

SUMMARY:
The goal of this clinical trial is to learn about the use of the Prone Positioner in pediatric patients with tracheostomies (trachs). The main question[s] it aims to answer are:

* What is the fit and satisfaction of the device?
* Does the device fulfill the goal of allowing infants with trachs participate in tummy time
* What aesthetic feedback will the study team receive on the prone positioner from families, therapists, and nursing staff.

Participants will be placed in the Prone Positioner, they will be monitored for their comfort/satisfaction with use, and how well they are able to be receive ventilation while in the device. Parents of these infants, as well as healthcare providers, will be surveyed on thoughts/suggestions for the Prone Positioner.

DETAILED DESCRIPTION:
A trained member of this study staff will be always present in the patient room during the fit test. For the fit test, a therapist from the study team will takes measurements of the infant and then place the infant in the prone positioner device. At no time will the baby be left alone or unsupported by staff. The study team will assess the physical fit, ease of getting the infant in and out of the device, and the patient's tolerance to being in the positioner.

Parents/guardians will be able to be present while the patient is in the device (if the parents are available and present at the time of fit testing) and immediately following the patient's removal from the device, the parents will be asked to complete a paper survey. The survey will ask for their perceptions of the device, initial reactions, and other qualitative data collected during the fit test. Healthcare providers who are not part of the study team will also be surveyed to obtain their thoughts/opinions on the device as well.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient infants located on the Pediatric Intensive Care Unit (PICU) or (Neonatal Intensive Care Unit (NICU) or being seen in the Vent clinic at Children's Mercy with tracheostomies between the ages of >44 weeks gestational age to 24 months of age with various size/weights of infants.
* Any race/ethnicity
* English speaker
* Males and females
* Caregivers
* Children's Mercy (CM) Occupational Therapists (OTs), Physical Therapists (PTs), Speech Therapists (STs) who have not seen the new prone positioner device.

Exclusion Criteria:

* Infants > 24 months of age
* Infants medically unstable as determined by attending physician in the PICU/NICU or Vent Clinic
* Infants with recent cardiac or abdominal surgery who have precautions or complications related to their surgery.
* Infants with weightbearing restrictions/fractures in their upper extremities.
* Non-English speakers * Wards of the state

Ages: 44 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Fit and Size of Prone Positioner | 45 minutes
  Evaluate the fit and size of the prone positioner prototype with infants with tracheostomies of varying ages/sizes

SECONDARY OUTCOMES:
Parental Satisfaction with Prone Positioner | Post patient use of positioner, survey to take a maximum of 10 minutes
  Evaluate if the prone positioner appeals to parents' satisfaction and trust in its use (i.e., does the device fulfill the goal of allowing infants with trachs participate in tummy time?)

OTHER OUTCOMES:
Improvement in Positioning Needs of Patients | Observed during the 45 min when patient is in Prone Positioner
  Evaluate if the current prone positioner design improves positioning needs of patients who have tracheostomies and are ventilator dependent
Aesthetic and Usability Feedback of Prone Positioner | Post patient use of positioner, survey to take a maximum of 10 minutes
  Gather aesthetic and usability feedback on the prone positioner from families, therapists, and nursing staff

CONTACTS AND LOCATIONS:
Overall Officials: Brandi Dorton, DPT, NTMTC, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) elements will only be made available to the study team within Children's Mercy Kansas City. These IPD will be protected to greatest extent possible by the study team through the use of encrypted files and password protected sign-ons.

REFERENCES:
- [Result] Hewitt L, Stanley RM, Okely AD. Correlates of tummy time in infants aged 0-12 months old: A systematic review. Infant Behav Dev. 2017 Nov;49:310-321. doi: 10.1016/j.infbeh.2017.10.001. Epub 2017 Nov 2. PMID 29096238
- [Result] Rocha NA, Tudella E. The influence of lying positions and postural control on hand-mouth and hand-hand behaviors in 0-4-month-old infants. Infant Behav Dev. 2008 Jan;31(1):107-14. doi: 10.1016/j.infbeh.2007.07.004. Epub 2007 Aug 17. PMID 17707512